CLINICAL TRIAL: NCT00411853
Title: An Open Phase II Clinical Trial of Fermented Wheat Germ Extract in Combination With Hormone Therapy for the Treatment of Hormone-Refractory Prostate Cancer Patients
Brief Title: Efficacy of FWGE in Combination With Hormone Therapy for the Treatment of Hormone-Refractory Prostate Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Rony Weitzen, Sheba Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-06-4232-RW-CTIL
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2009-07-31 (Estimated); Status verified 2009-07

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: Prostate, Hormone Refractory, Cancer
MeSH Terms: conditions — Neoplasms | interventions — Avemar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fermented Wheat germ extract — Fermented Wheat Germ powder, given orally, per os, 17 gram daily

SUMMARY:
We propose in this study to treat hormone refractory prostate cancer (HRPC) patients., with a novel preparation of fermented wheat germ nutriment (FWGE), in combination with the 1st line hormone therapy, the gonadotropin releasing hormone (GnRH), which stopped being effective. The study will be conducted during two years with 60 patients. The efficacy will be assessed in terms of clinical and serological response and by specific questionnaires.

This concept is based on previous reports regarding other diseases such as colon cancer, where the addition of a new drug to a drug which previously had failed, improved the patients' survival, the quality of life and the clinical parameters. In addition, preclinical data have shown activity of that regimen in prostate cancer cell lines and in animals' models.

FWGE exhibits a wide variety of mode of actions, in a wide range of malignant tumors. It increased the natural immune responses while decreasing the systemic inflammation often present in cancer patients. It reduced the growth of human prostate tumor xenograft in mice and prolonged their survival. It delayed disease progression, increased overall survivals, improve quality of life and reduce oxidative stress.

The long-term goal of this research is that the addition of FWGE to a drug which previously had failed, would slow down disease progression in patients with advanced and thus refractory cancers, improving the patients' quality of life, their clinical parameters and survival.

DETAILED DESCRIPTION:
Background and Significance

1. The challenge:

   Prostate cancer is a major worldwide health problem and is the most frequently diagnosed malignancy in men today. In the United States prostate cancer is the most common malignancy found in men accounting for more than 29% of all diagnosed cancer and approximately 13% of all cancer deaths. Nearly one in six men will be diagnosed with the disease at some time in their lives. In 2003 alone, an estimated 221,000 men in the United States were diagnosed with prostate cancer. In 1999, 37,000 deaths were attributed to prostate cancer in the United States, and in 2003 more than 28,000 died of the disease. Hormone-refractory prostate cancer (HRPC) is one of the most aggressive cancers. It is the second ranking cause of cancer-related deaths. Patients with localized disease have the option of radiation therapy or radical prostatectomy as definitive treatment modalities for curing the disease. However the cancer recurs in its metastatic form in 20-30% of these patients. In addition, approximately 10 % of patients diagnosed with the disease already have distant metastases, making localized therapy irrelevant. The primary treatment for the advanced state of prostate cancer is androgen deprivation therapy, to inhibit the testosterone production that facilitates prostate tumor growth. Androgen deprivation therapy is administered either by surgical castration or by medications that block testosterone production. While this treatment is effective in 85%-95% of patients, the response time lasts approximately for 12 -24 months, after which the cancer progresses to its androgen-insensitive stage. The androgen independent prostate cancer cells progress to metastatic disease. Limited treatment options exist for the hormone refractory prostate cancer (HRPC) patient, and median survival time rarely exceeds one year.

   Once androgen independence has occurred, conventional chemotherapy for the treatment of metastatic cancer has shown limited activity in patients in addition to causing toxic side effects. While new chemotherapeutic regimens and hormonal agents are being tested, the survival and quality of life of these HRPC patients remains low.
2. The innovation:

We propose to treat progressing HRPC patients with a novel combination of 1st line of hormone therapy (GnRH analogues) with the non-toxic dietary supplement fermented wheat germ nutriment (FWGE). This suggestion is based on preclinical data showing activity of the regimen in prostate cancer cell lines and in animal models. Furthermore, there are previous reports regarding other diseases such as colon cancer, where the addition of a new treatment to a therapy which had previously failed, improved patient survival, quality of life and the clinical parameters.

The characteristics of Fermented wheat germ extract (FWGE) Fermented wheat germ extract with a standardized complex mixture of molecules is termed FWGE. The product is manufactured under GMP conditions, and is available as a water-soluble granulate, which administered orally.

The compound is approved as a medical food for cancer patients. It has been recently classified in the US as GRAS (Generally Recognized as Safe), and is used for complementing the standard anticancer treatments.

The molecular targets of FWGE include poly (ADP-ribose) polymerase (PARP), major histocompatibility complex (MHC) class I, transketolase (TK), ribonucleotide reductase (RNR) and, intracellular adhesion molecule (ICAM) 1. By activating the caspase-3 downstream proteases, FWGE treatment results in cleavage of PARP thus, preventing DNA repair in cancer cells.

FWGE treatment decreases major histocompatibility complex class I (MHC-I) in cancer cells. MHC-I down regulation in cancer cells leads to an increased natural killer (NK) cells' activity. NK cells are considered as the first line of anticancer immune defense.

TK is the key enzyme of the reductive pentose cycle. In cancer cells this cycle is responsible for supplying these cells' increased need for ribose molecules necessary for synthesis the sugar chains of the nucleic acids. RNR enzymes, which are strongly inhibited by FWGE, catalyze the synthesis of the DNA components.

It has been known that a tumor can not grow bigger than 2 mm in diameter except if it is able to synthesize its own blood vessels (angiogenesis process). The blood vessels in tumors lack the protein ICAM-1, which is responsible for facilitating the transfer of anticancer immune cells (e. g. macrophages) via the vessels' walls into the tumor. FWGE treatment increases the synthesis of ICAM-1.

In addition, FWGE has a wide therapeutic window: In order to observe any toxicity (effects on normal cells), more than 50 times higher dosage of FWGE than the recommended one for therapy is needed. This very positive toxicity profile gives a wide therapeutic window for the applicability of this product.

Recently, it has also been shown that FWGE is a strong but, non-selective inhibitor of the cyclooxygenases 1 and 2 thus, this preparation has an anti-inflammatory activity.

The preparation has also been shown to induce apoptosis in gastric carcinoma cells.

Advantages of FWGE:

* The FWGE preparation is non-toxic and safe. This serves as a major consideration in its selection for the treatment of advanced cancer patients who suffer from low performance status and consequently have a poor quality of life.
* FWGE is orally administrated.
* The FWGE preparation exhibits a wide variety of mode of actions, in a wide range of malignant tumors.
* The product is able to increase the natural immune responses, while decreasing the systemic inflammation often present in the patients.
* It is anticipated that FWGE, by complementing therapeutic efficacy of the standard hormonal anticancer treatments, could suppress disease progression, thus prolonging patients' survival and improving quality of life parameters.

ELIGIBILITY:
Subject Inclusion Criteria:

1. Age >18
2. Histology/cytology diagnosis of prostate cancer
3. Measurable disease as identified by tumor imaging (e.g. CT, MRI) or PSA values greater than 1.5 ng/ml, and rising in 3 consecutive measurements.
4. failure of 1st line hormone therapy (GnRH analogues)
5. ECOG performance status 0-2

Subject Exclusion Criteria:

1. Concurrent use of systemic anti-neoplastic therapy
2. Patients who had received systemic chemotherapy for prostate cancer.
3. Patients receiving an investigational agent within the past 30 days of study entry.
4. Patients with evidence of circumstances that are likely to interfere with the absorption of orally administrated products.
5. patients with co-morbidities considered to potentially influence the outcome of treatment in the judgment of the investigator (life-threatening diseases such as heart failure)
6. ECOG performance status > 2

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-06; Primary Completion 2011-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Response rate in 16 weeks. | 1 year

SECONDARY OUTCOMES:
Quality of life in 16 weeks | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rony Weitzen, MD, Principal Investigator — Oncology Division Sheba Medical Center
Locations (1):
- Oncology Division Sheba Medical Center, Tel Litwinsky, Ramat Gan, Israel

REFERENCES:
- [Derived] Weitzen R, Epstein N, Oberman B, Shevetz R, Hidvegi M, Berger R. Fermented Wheat Germ Extract (FWGE) as a Treatment Additive for Castration-Resistant Prostate Cancer: A Pilot Clinical Trial. Nutr Cancer. 2022;74(4):1338-1346. doi: 10.1080/01635581.2021.1952457. Epub 2021 Jul 21. PMID 34286638